CLINICAL TRIAL: NCT00111969
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Assess the Effects of the Celacade™ System on Mortality and Morbidity in Patients With Chronic Heart Failure
Brief Title: ACCLAIM - Advanced Chronic Heart Failure CLinical Assessment of Immune Modulation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vasogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0202; NCT00386295 (obsolete NCT alias)
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Heart Failure, Congestive
Keywords: Heart failure; Immune modulation therapy; Inflammation; Chronic systolic heart failure
MeSH Terms: conditions — Heart Failure; Inflammation

INTERVENTIONS:
Device: Celacade™ system

SUMMARY:
The purpose of this study is to test the safety and efficacy of the Celacade™ system in reducing the risk of mortality and cardiovascular hospitalizations in patients with chronic systolic heart failure.

DETAILED DESCRIPTION:
Evidence continues to accumulate on the importance of inflammation in the development and progression of heart failure (HF). The Celacade™ system may reduce chronic inflammation by stimulating the immune system's physiological anti-inflammatory response. The ACCLAIM study is an international, approximately 2,000-patient, Phase III clinical research study designed to test the safety and efficacy of the Celacade™ system in reducing the risk of mortality and cardiovascular hospitalizations in patients with chronic systolic HF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older.
* New York Heart Association (NYHA) Class II to IV.
* Left ventricular ejection fraction (LVEF) ≦ 30%, measured within the past six months (by any technique), unless there was a cardiovascular event that could have modified the LVEF during that period (e.g., coronary artery bypass grafting [CABG], myocardial infarction [MI]). If the patient was started on a beta-blocker or biventricular pacing (cardiac resynchronization therapy, or CRT), the LVEF measurement must have been at least three months after starting the therapy.
* Hospitalized for heart failure; OR, received intravenous (IV) administration of an inotropic agent (therapeutic dose for HF), human B-natriuretic peptide, or IV diuretic (minimum 40 mg of furosemide or equivalent) in a clinic, outpatient or emergency department within the past 12 months (stable for at least 2 weeks). Exceptions: patients in NYHA Class III or IV who have a LVEF of < 25%.
* On standard therapy for congestive heart failure (CHF), which must include angiotensin converting enzyme (ACE) inhibitors or angiotensin II receptor blocker (ARB) (unless contraindicated or patient is intolerant), with or without other appropriate agents. If on a beta-blocker, patient must have been on a beta-blocker for at least three months.
* No changes in active cardiac medications for heart failure during the two weeks prior to randomization.
* Written informed consent

Exclusion Criteria:

* Inability to comply with the conditions of the protocol.
* Presence of a transplanted tissue or organ or left ventricular assist device (LVAD) (or the expectation of the same within the next 12 months).
* Planned Automatic Implantable Cardiac Defibrillator (AICD) or CRT within the next 12 months.
* Acute MI, or CABG, percutaneous coronary intervention (PCI), AICD, or CRT within the past three months.
* Need for chronic intermittent inotropic therapy.
* Malignancy: evidence of disease within the previous five years. Exceptions: basal cell carcinoma, provided that it is neither infiltrating nor sclerosing, and carcinoma in situ of the cervix.
* Active myocarditis or early postpartum cardiomyopathy (within the first six months of delivery).
* Systemic corticosteroids, cytostatics, immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), and DNA depleting or cytotoxic drugs taken within four weeks prior to study treatment.
* Pregnancy, or patients of childbearing potential not using adequate contraceptive methods.
* Porphyria.
* Allergy to sodium citrate or any "caine" type of local anesthetic.
* Previous Celacade™ treatment.
* Patient scheduled for hospice care.
* Clinically relevant abnormal findings in the clinical history, physical examination, electrocardiogram (ECG), or laboratory tests at the screening assessment that would interfere with the objectives of the study or that would, in the investigator's opinion, preclude safe completion of the study. Abnormal findings could include: known HIV infection or other immunodeficiency state, chronic active viral infection (such as hepatitis B or C), acute systemic infections (defined as patients undergoing treatment with antibiotics), gastrointestinal tract bleeding, or any severe or acute concomitant illness or injury.
* Any other medical, social, or geographical factor that would make it unlikely that the patient could comply with study procedures (e.g., alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or a history of noncompliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2016
Dates: Start 2003-06; Study Completion 2005-11

PRIMARY OUTCOMES:
Mortality
Cardiovascular hospitalization

SECONDARY OUTCOMES:
Clinical status
Health-related patient quality
Healthcare resource utilization

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Parker, PhD, Study Director — Vasogen Inc.

REFERENCES:
- [Derived] Torre-Amione G, Anker SD, Bourge RC, Colucci WS, Greenberg BH, Hildebrandt P, Keren A, Motro M, Moye LA, Otterstad JE, Pratt CM, Ponikowski P, Rouleau JL, Sestier F, Winkelmann BR, Young JB; Advanced Chronic Heart Failure CLinical Assessment of Immune Modulation Therapy Investigators. Results of a non-specific immunomodulation therapy in chronic heart failure (ACCLAIM trial): a placebo-controlled randomised trial. Lancet. 2008 Jan 19;371(9608):228-36. doi: 10.1016/S0140-6736(08)60134-8. PMID 18207018
- See also: Related Info — http://www.vasogen.com